CLINICAL TRIAL: NCT04839913
Title: Seroprevalence of SARS-CoV-2 in Unselected Surgical Patients: an Update From an Unicentric, Regional Study
Brief Title: Seroprevalence of SARS-CoV-2 in Unselected Surgical Patients: an Unicentric, Regional Study
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Fabio Medas, Surgical researcher, University of Cagliari
Other Study IDs: COVID-SER
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV Infection; Seroprevalence; Covid19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Antibodies testing — Serologic test for both SARS-COV-2 IgG and IgM

SUMMARY:
The investigator analyzed the data of the patients admitted to the surgical department during the period 1St September - 10Th December 2020 to estimate the seroprevalence of SARS-CoV-2 infection in the setting of a non-dedicated COVID-19 hospital and in a mild CoV-2 incidence area and to evaluate the difference of seroprevalence between Spring and Fall seasons in a cohort of patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to our unit who had performed SARS-COV-2 serologic test

Exclusion Criteria:

* age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a cohort of elective surgical patients admitted to our unit in the 2020 fall period
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
SARS-COV-2 seroprevalence | 1St September - 10Th December 2020
  SARS-COV-2 IgG and IgM seroprevalence between spring and fall period

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No